CLINICAL TRIAL: NCT02448173
Title: A Randomized Multicenter Study of Active Specific Immunotherapy With OncoVax® in Patients With Stage II Colon Cancer
Brief Title: A Multicenter Study of Active Specific Immunotherapy With OncoVax® in Patients With Stage II Colon Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vaccinogen Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI-2005-04
Record Dates: First submitted 2015-05-06; First posted 2015-05-19 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Stage II Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OncoVAX and Surgery (Experimental): Autologous Specific Immunotherapy given intradermally following surgical resection of Stage II colon cancer
  Interventions: Biological: OncoVAX and Surgery; Procedure: Surgery
- Surgery (Active Comparator): Surgical resection of Stage II colon cancer
  Interventions: Procedure: Surgery

INTERVENTIONS:
Biological: OncoVAX and Surgery — OncoVAX is comprised of sterile, live but non-dividing tumor cells obtained following standard-of-care surgical tumor resection for Stage II colon cancer
  Arms: OncoVAX and Surgery
Procedure: Surgery — Surgical resection of Stage II colon cancer

SUMMARY:
OncoVAX® is the first cancer therapy that both prevents cancer recurrence and

addresses the diversity of cancer cells. In this pivotal randomized, multicenter Phase

IIIb study in patients with Stage II colon cancer, OncoVAX is designed to use a patient's

own cancer cells to mobilize the body's immune system to prevent the return of colon

cancer following surgery.

DETAILED DESCRIPTION:
OncoVAX is an active specific immunotherapeutic (ASI) stimulating a patient's immune

response to autologous (patient-specific) tumor cells. It is comprised of sterile, live but

non-dividing tumor cells obtained following standard-of-care surgical tumor resection for

Stage II colon cancer. Within 35 days following surgery, patients are immunized with

OncoVAX to prevent disease recurrence, which is incurable and occurs in up to 35% of

patients. Patients are given three injections once per week for three weeks, followed

by a booster shot after six months. A previously completed Phase III trial

published in The Lancet showed that OncoVAX cut the risk of recurrence by 61% in

patients with Stage II colon cancer. The primary endpoint is Disease-Free Survival:

defined as the time from curative surgery to the objective test confirming tumor

recurrence or death due to any cause. The secondary endpoints are Overall Survival

and Recurrence-Free-Interval. An interim analysis will be performed at a significance

level of 0.005 once 2/3 of anticipated events have occurred, resulting in a significance

level of 0.0483 at the end of the study. A total of 550 patients is planned, randomized

1:1 to receive OncoVAX® plus surgery (n=275) or surgery alone (n=275).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage II (IIA = T3N0M0, IIB = T4aN0M0, IIC = T4bN0M0) disease.
* Patients must have undergone curative resection and have no evidence of residual or metastatic disease.
* Following curative resection patients must have a CEA within normal limits. If elevated prior to resection, it must return to normal within 21 days post surgery and prior to randomization.

Exclusion Criteria:

* Patients with prior radiation therapy or chemotherapy or a prior malignancy of any type will be excluded. However, subjects with prior, curatively-treated squamous cell or basal cell carcinoma of the skin or carcinoma in situ of the cervix will be eligible for participation in this study.
* Patients with more than one malignant primary colon cancer will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2031-08 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | Up to Five years
  Defined as time from randomization to the date of the first objective test confirming tumor recurrence or death due to any cause

SECONDARY OUTCOMES:
Overall Survival | Up to Five Years
  Defined as the time from randomization to death due to any cause
Recurrence-Free Interval | Up to Five Years
  Defined as the time from randomization to the first objective test confirming tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Hanna, Jr, PhD, Study Chair — Vaccinogen Inc; Herbert C. Hoover, MD, Study Director — Vaccinogen Inc
Locations (1):
- Halifax Health Medical Center, Port Orange, Florida, United States